CLINICAL TRIAL: NCT02884466
Title: Comparison of Two Multidisciplinary Rehabilitation Interventions in Patients With Chronic Low Back Pain - A Randomised Controlled Clinical Trial
Brief Title: Comparison of Two Multidisciplinary Rehabilitation Interventions in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Sano 1
Record Dates: First submitted 2016-08-19; First posted 2016-08-31 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive a multidisciplinary rehabilitation intervention consisting of: 1) a pre-admission day, 2) two weeks of home-based activities, 3) two-week inpatient period, 4) four weeks of home-based activities, 5) 1st two-days inpatient follow-up, 6) six weeks of home-based activities and 7) 2nd two-days inpatient follow-up.
  Interventions: Behavioral: Multidisciplinary rehabilitation intervention
- Usual care group (Active Comparator): The usual care group will receive a four-week inpatient multidisciplinary rehabilitation intervention.
  Interventions: Behavioral: Multidisciplinary rehabilitation intervention

INTERVENTIONS:
Behavioral: Multidisciplinary rehabilitation intervention — Both groups will receive examination and medicine adjustment from a rheumatologist, and treatment from physiotherapist, occupational therapist and nursing staff, respectively. The multidisciplinary rehabilitation intervention in both groups will be based on the biopsychosocial model of illness. The inpatient stays of 8-10 hours per day will consist of 1) group tuition, 2) group and individual treatment and 3) unassisted training sessions.

SUMMARY:
Introduction Chronic low back pain (CLBP) is a highly prevalent health condition, and the leading cause of years lived with disability. The high prevalence causes a substantial impact on patients, communities and health-care systems. There is a continuing challenge to offer evidence-based rehabilitation for patients with CLBP. There is a lack of studies on adequate follow-up approaches to maintain successful treatment. No earlier study has assessed if the positive treatment effects of a multidisciplinary rehabilitation intervention can be maintained with an intervention alternating between inpatient interventions and home-based activities.

Aim To assess if a novel multidisciplinary rehabilitation intervention is more effective in maintaining successful treatment after 6 months, than a usual multidisciplinary rehabilitation intervention in patients with CLBP.

The novel intervention is a 14-week program alternating between in total three weeks of inpatient intervention and home-based activities. This alternation allows the participants time and opportunity to adapt and transfer inpatient learning to activities and participation in their own environment in interaction with everyday life situations and surroundings. Usual care is a four-week inpatient intervention. It is hypothesized that the intervention will be superior to usual care.

Method The study will be conducted at The Danish Rheumatism Associations' rehabilitation centre Sano Aarhus. 160 participants with CLBP will be randomly allocated to one of two groups. The novel intervention consists of: 1) a pre-admission day, 2) two weeks of home-based activities, 3) two-week inpatient period, 4) four weeks of home-based activities, 5) 1st two-days inpatient follow-up, 6) six weeks of home-based activities and 7) 2nd two-days inpatient follow-up. Usual care consists of a four-week inpatient intervention.

The two groups will be compared according to disability, pain, pain self-efficacy, quality of life, depression and exercise capacity.

Relevance The present study has emerged out of the fields where patients, clinicians and researchers intersect and is consequently highly clinically relevant. If positive treatment effects can be maintained or even improved in the long term, the results may serve as inspiration for the design of multidisciplinary rehabilitation interventions in clinical practice; this will be valuable for future patients with CLBP.

DETAILED DESCRIPTION:
Introduction Chronic low back pain (CLBP) is a highly prevalent health condition, and the leading cause of years lived with disability both globally and in Denmark. In the majority of patients with CLBP, no underlying pathology or cause can be identified and CLBP is acknowledged to be multifactorial.

CLBP is defined by symptoms lasting for a period longer than three months. The high prevalence of CLBP causes a substantial impact on patients and their families, communities and health-care systems, as well as a financial burden. Besides pain and disability people with CLBP often experience psychosocial consequences with signs of anxiety and depression and effects on social, leisure, and work life. Recognition of the physical, psychological and social consequences of CLBP led to the development of the widely accepted biopsychosocial model in the understanding and managing of CLBP.

The World Health Organization's (WHO) International Classification of Functioning, Disability and Health (ICF) provides a framework for applying the biopsychosocial model into clinical practice, especially into rehabilitation. By emphasizing, that disability is a dynamic interaction between the dimensions of body function, activity, participation, and environmental and personal factors, ICF helps treating the patients rather than only their low back pain by addressing all the biopsychosocial dimensions of their disability.

Disability itself arises through complex and multi-factorial mechanisms and therefore, rehabilitation processes are defined as complex health interventions undertaken in a complex environment. Rehabilitation is rather a process than a treatment or specific action, and a multidisciplinary team most effectively manages the complex problems seen in rehabilitation. Rehabilitation has many potential active ingredients, and combining the different components in a whole is more than the sum of its parts.

There is a continuing challenge to offer evidence-based rehabilitation for patients with CLBP. A systematic review by Kamper identified and assessed risk of bias in 12 randomized controlled trials (RCT's) comparing two multidisciplinary rehabilitation interventions. In March 2016 we performed an updated literature search in PubMed identical to that of the review and identified one additional RCT comparing two multidisciplinary interventions. Risk of bias in the additional study was assessed using Cochrane risk of bias tool (The Cochrane Collaboration ) identical to the review.

Nine of the 13 studies had disability and pain as primary or secondary outcome. The multidisciplinary interventions being compared varied across the nine studies in content and/or time frame. As the studies were very heterogenic, a pooled comparison and description was not possible. Overall the nine studies showed that multidisciplinary rehabilitation had a positive effect on disability and pain in the short and medium term, but there were discrepancy in the studies whether the effect can be maintained in the long term. A literature search identified two studies on follow-up care. One study tested the effect of multidisciplinary rehabilitation with subsequent booster sessions conducted by telephone within 12 months after discharge, and found only slight advantages, but no statistical significance of the booster sessions. The other study compared a 3-month exercise follow-up program and routine follow-up on patients with CLBP who had completed a 3-week outpatient multidisciplinary rehabilitation program. Favourable outcomes after one year were observed in both groups, but only patients attending the exercise follow-up program improved in disability.

There is a lack of studies on adequate follow-up approaches to maintain successful treatment. No earlier study has assessed if the positive treatment effects of a multidisciplinary rehabilitation intervention can be maintained with an intervention alternating between inpatient interventions and home-based activities.

Aim To assess if a novel multidisciplinary rehabilitation intervention is more effective in maintaining successful treatment after 6 months, than a usual multidisciplinary rehabilitation intervention in patients with chronic low back pain.

The novel intervention is a 14-week program alternating between in total three weeks of inpatient intervention and home-based activities. This alternation will allow the participants time and opportunity to adapt and transfer inpatient learning to activities and participation in their own environment in interaction with everyday life situations and surroundings. Furthermore, the novel intervention will consist of a higher degree of patient involvement than the usual intervention. Usual care is a four-week inpatient intervention.

Objectives (i) To compare changes in the two multidisciplinary rehabilitation groups on disability, pain, pain self-efficacy, quality of life, anxiety/depression and exercise capacity.

(ii) To examine the association between changes in disability versus changes in pain, pain self-efficacy, quality of life, anxiety/depression and exercise capacity.

Hypotheses (i) The intervention group will experience a five points larger improvement in Oswestry Disability Index compared to usual care. Furthermore, the intervention group will experience a larger improvement in pain, pain self-efficacy, quality of life, anxiety/depression and exercise capacity compared to usual care.

(ii) There is negative association between changes in disability and quality of life, pain self-efficacy and exercise capacity, respectively. There is a positive association between disability and pain and anxiety/depression, respectively. The strongest association will be between disability and pain self-efficacy.

Materials and methods Study setting All participants will be recruited from, treated and tested at Sano Aarhus, Denmark. A rheumatologist will perform the selection of participants based on the clinical problem of referral.

Randomization An independent administrative assistant will perform a randomly allocated computer-generated randomization of participants into either intervention or control group. Stratified randomization on the basis of Oswestry Disability Index score below and above 40 will be used in order to achieve approximate balance of disability in the two groups. 1:1 allocation in blocks of 6 will be used. Due to waiting time, randomization will take place in average 5-6 months before study start.

Blinding As both interventions will be performed in the same physical setting at the same time, blinding of participants and intervening clinicians will not be possible due to knowledge of content and duration of the intervention the participants are allocated to. Intervening clinicians involved in the treatment of both groups will assess physical status of the participants. In order to raise equal expectations, participants will be blinded to the study hypothesis by telling them the RCT is intended to compare two equal multidisciplinary rehabilitation interventions both meeting current scientific standards and appropriate to improve health status.

The researchers involved in the statistical analyses will be blinded to treatment groups.

Sample size Oswestry Disability Index was used for sample size calculation. Based on data from the literature and a pilot study on 25 patients with CLBP from Sano, mean change is estimated to 10 in the intervention group and 5 in the control group, and the standard deviation on the changes is estimated to 10. Using 80% power and a significance level of 0.05, 64 participants will be required in each group. A dropout rate of 20% is estimated, for what reason it will be planned to recruit a total of 160 participants.

Interventions The content of both interventions will be described in details in a study protocol as recommended for complex interventions.

Both groups will be managed by the same multidisciplinary staff in the same physical setting at the same time. Participants in the two groups will inevitably meet each other, and thus both they and the multidisciplinary staff will have the opportunity to compare and discuss the different rehabilitation interventions. Despite the possible overflow between the two rehabilitation interventions, the present parallel design has been preferred rather than a staggered design where waiting time and external circumstances would have been different between the two groups.

Data collection Demographics and PROMs will be collected before the randomization (baseline), and due to 5-6 months of waiting time again at the beginning of the inpatient rehabilitation intervention (intervention start). Exercise capacity test performed by a trained physiotherapist using a standardized protocol, and clinical and neurological findings collected by an experienced rheumatologist using a standardized examination protocol, will be collected at the first inpatient contact.

Follow-up data will be collected at the end of the inpatient rehabilitation intervention, at each follow-up (intervention group) and at 6 and 12 months. Participants dropping out will be asked to fill in the PROMs at 6 months.

Participants enter data directly in a database via a link. In order to minimize missing data a reminder will be send via email after one week. If participants are unable to fill out the electronic versions, an independent administrative assistant will enter data from a paper copy of the questionnaires.

Perspective The present study has emerged out of the fields where patients, clinicians and researchers intersect and is consequently highly clinically relevant. If positive treatment effects can be maintained or even improved in the long term, the results may serve as inspiration for the design of multidisciplinary rehabilitation interventions in clinical practice; this will be valuable for future patients with CLBP.

ELIGIBILITY:
Inclusion Criteria:

* low back pain for more than 12 months with or without sciatica and/or with or without generalized pain identified by ICD-10 codes
* Oswestry Disability score > 20.

Exclusion Criteria:

* a rated physical status of > 3 according to the American Society of Anesthesiologists Physical Status Classification System
* axial spondyloarthritis
* spinal fracture within the last 3 months
* severe osteoporosis
* active cancer
* active psychiatric pathology assessed by general practitioner before referral
* pregnancy
* low Danish language skills.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2016-10; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
The Oswestry Disability Index | 28 months

SECONDARY OUTCOMES:
Numerical Rating Scale | 28 months
The Pain Self-Efficacy Questionnaire | 28 months
EQ-5D | 28 months
Major Depression Inventory | 28 months
Aastrands cycle test | 28 months
Three questions on physical activity | 28 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Mette Schmidt, MSc, Principal Investigator — Sano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Global Burden of Disease Study 2013 Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 301 acute and chronic diseases and injuries in 188 countries, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Aug 22;386(9995):743-800. doi: 10.1016/S0140-6736(15)60692-4. Epub 2015 Jun 7. PMID 26063472
- [Background] Hoy D, Brooks P, Blyth F, Buchbinder R. The Epidemiology of low back pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):769-81. doi: 10.1016/j.berh.2010.10.002. PMID 21665125
- [Background] Driscoll T, Jacklyn G, Orchard J, Passmore E, Vos T, Freedman G, Lim S, Punnett L. The global burden of occupationally related low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):975-81. doi: 10.1136/annrheumdis-2013-204631. Epub 2014 Mar 24. PMID 24665117
- [Background] Statens Institut for Folkesundhed. Folkesundhedsrapporten, Danmark 2007 Kapitel 7. Muskel- og skeletsygdomme. Available at: http://www.si-folkesundhed.dk/upload/kap_7_muskel-_og_skeletsygdomme.pdf. Accessed 03/29, 2016.
- [Background] Waddell G. Chapter 6. Risk factors for back pain. The Back Pain Revolution. 2nd ed ed. London: Elsevier Limited: Churchill Livingstone; 2004. p. 91.
- [Background] Kamper SJ, Apeldoorn AT, Chiarotto A, Smeets RJ, Ostelo RW, Guzman J, van Tulder MW. Multidisciplinary biopsychosocial rehabilitation for chronic low back pain: Cochrane systematic review and meta-analysis. BMJ. 2015 Feb 18;350:h444. doi: 10.1136/bmj.h444. PMID 25694111
- [Background] Hoy D, March L, Brooks P, Blyth F, Woolf A, Bain C, Williams G, Smith E, Vos T, Barendregt J, Murray C, Burstein R, Buchbinder R. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):968-74. doi: 10.1136/annrheumdis-2013-204428. Epub 2014 Mar 24. PMID 24665116
- [Background] Waddell G. Chapter 5. The epidemiology of back pain. The Back Pain revolution London: Elsevier Limited: Churchill Livingstone; 2004. p. 71.
- [Background] Chiarotto A, Deyo RA, Terwee CB, Boers M, Buchbinder R, Corbin TP, Costa LO, Foster NE, Grotle M, Koes BW, Kovacs FM, Lin CW, Maher CG, Pearson AM, Peul WC, Schoene ML, Turk DC, van Tulder MW, Ostelo RW. Core outcome domains for clinical trials in non-specific low back pain. Eur Spine J. 2015 Jun;24(6):1127-42. doi: 10.1007/s00586-015-3892-3. Epub 2015 Apr 5. PMID 25841358
- [Background] Wade D. Rehabilitation - a new approach. Part two: the underlying theories. Clin Rehabil. 2015 Dec;29(12):1145-54. doi: 10.1177/0269215515601175. PMID 26581670
- [Background] Pincus T, Kent P, Bronfort G, Loisel P, Pransky G, Hartvigsen J. Twenty-five years with the biopsychosocial model of low back pain-is it time to celebrate? A report from the twelfth international forum for primary care research on low back pain. Spine (Phila Pa 1976). 2013 Nov 15;38(24):2118-23. doi: 10.1097/BRS.0b013e3182a8c5d6. PMID 23970112
- [Background] Waddell G. Chapter 14. The biopsychosocial model. The Back Pain Revolution. 2nd ed ed. London: Elsevier Limited: Churchill Livingstone; 2004. p. 265.
- [Background] Wade DT, Smeets RJ, Verbunt JA. Research in rehabilitation medicine: methodological challenges. J Clin Epidemiol. 2010 Jul;63(7):699-704. doi: 10.1016/j.jclinepi.2009.07.010. Epub 2009 Sep 27. PMID 19788953
- [Background] Wade D. Rehabilitation - a new approach. Part three: the implications of the theories. Clin Rehabil. 2016 Jan;30(1):3-10. doi: 10.1177/0269215515601176. PMID 26659136
- [Background] Momsen AM, Rasmussen JO, Nielsen CV, Iversen MD, Lund H. Multidisciplinary team care in rehabilitation: an overview of reviews. J Rehabil Med. 2012 Nov;44(11):901-12. doi: 10.2340/16501977-1040. PMID 23026978
- [Background] Oakley A, Strange V, Bonell C, Allen E, Stephenson J; RIPPLE Study Team. Process evaluation in randomised controlled trials of complex interventions. BMJ. 2006 Feb 18;332(7538):413-6. doi: 10.1136/bmj.332.7538.413. PMID 16484270
- [Background] Hart T, Bagiella E. Design and implementation of clinical trials in rehabilitation research. Arch Phys Med Rehabil. 2012 Aug;93(8 Suppl):S117-26. doi: 10.1016/j.apmr.2011.11.039. PMID 22840878
- [Background] Mangels M, Schwarz S, Worringen U, Holme M, Rief W. Evaluation of a behavioral-medical inpatient rehabilitation treatment including booster sessions: a randomized controlled study. Clin J Pain. 2009 Jun;25(5):356-64. doi: 10.1097/AJP.0b013e3181925791. PMID 19454868
- [Background] Abbasi M, Dehghani M, Keefe FJ, Jafari H, Behtash H, Shams J. Spouse-assisted training in pain coping skills and the outcome of multidisciplinary pain management for chronic low back pain treatment: a 1-year randomized controlled trial. Eur J Pain. 2012 Aug;16(7):1033-43. doi: 10.1002/j.1532-2149.2011.00097.x. Epub 2012 Jan 19. PMID 22337646
- [Background] Bendix AE, Bendix T, Haestrup C, Busch E. A prospective, randomized 5-year follow-up study of functional restoration in chronic low back pain patients. Eur Spine J. 1998;7(2):111-9. doi: 10.1007/s005860050040. PMID 9629934
- [Background] Harkapaa K, Jarvikoski A, Mellin G, Hurri H. A controlled study on the outcome of inpatient and outpatient treatment of low back pain. Part I. Pain, disability, compliance, and reported treatment benefits three months after treatment. Scand J Rehabil Med. 1989;21(2):81-9. PMID 2526364
- [Background] Leeuw M, Goossens MEJB, van Breukelen GJP, de Jong JR, Heuts PHTG, Smeets RJEM, Koke AJA, Vlaeyen JWS. Exposure in vivo versus operant graded activity in chronic low back pain patients: results of a randomized controlled trial. Pain. 2008 Aug 15;138(1):192-207. doi: 10.1016/j.pain.2007.12.009. Epub 2008 Feb 1. PMID 18242858
- [Background] Linton SJ, Boersma K, Jansson M, Svard L, Botvalde M. The effects of cognitive-behavioral and physical therapy preventive interventions on pain-related sick leave: a randomized controlled trial. Clin J Pain. 2005 Mar-Apr;21(2):109-19. doi: 10.1097/00002508-200503000-00001. PMID 15722803
- [Background] Nicholas MK, Wilson PH, Goyen J. Operant-behavioural and cognitive-behavioural treatment for chronic low back pain. Behav Res Ther. 1991;29(3):225-38. doi: 10.1016/0005-7967(91)90112-g. PMID 1831972
- [Background] Smeets RJEM, Vlaeyen JWS, Hidding A, Kester ADM, van der Heijden GJMG, Knottnerus AJ. Chronic low back pain: physical training, graded activity with problem solving training, or both? The one-year post-treatment results of a randomized controlled trial. Pain. 2008 Feb;134(3):263-276. doi: 10.1016/j.pain.2007.04.021. Epub 2007 May 10. PMID 17498879
- [Background] Kole-Snijders AM, Vlaeyen JW, Goossens ME, Rutten-van Molken MP, Heuts PH, van Breukelen G, van Eek H. Chronic low-back pain: what does cognitive coping skills training add to operant behavioral treatment? Results of a randomized clinical trial. J Consult Clin Psychol. 1999 Dec;67(6):931-44. doi: 10.1037//0022-006x.67.6.931. PMID 10596514
- [Background] Meng K, Seekatz B, Roband H, Worringen U, Vogel H, Faller H. Intermediate and long-term effects of a standardized back school for inpatient orthopedic rehabilitation on illness knowledge and self-management behaviors: a randomized controlled trial. Clin J Pain. 2011 Mar-Apr;27(3):248-57. doi: 10.1097/AJP.0b013e3181ffbfaf. PMID 21178600
- [Background] Skouen JS, Grasdal AL, Haldorsen EM, Ursin H. Relative cost-effectiveness of extensive and light multidisciplinary treatment programs versus treatment as usual for patients with chronic low back pain on long-term sick leave: randomized controlled study. Spine (Phila Pa 1976). 2002 May 1;27(9):901-9; discussion 909-10. doi: 10.1097/00007632-200205010-00002. PMID 11979157
- [Background] van den Hout JH, Vlaeyen JW, Heuts PH, Zijlema JH, Wijnen JA. Secondary prevention of work-related disability in nonspecific low back pain: does problem-solving therapy help? A randomized clinical trial. Clin J Pain. 2003 Mar-Apr;19(2):87-96. doi: 10.1097/00002508-200303000-00003. PMID 12616178
- [Background] Linden M, Scherbe S, Cicholas B. Randomized controlled trial on the effectiveness of cognitive behavior group therapy in chronic back pain patients. J Back Musculoskelet Rehabil. 2014;27(4):563-8. doi: 10.3233/BMR-140518. PMID 25096315
- [Background] The Cochrane Collaboration. The Cochrane Collaboration's tool for assessing risk of bias. Available at: http://handbook.cochrane.org/chapter_8/table_8_5_a_the_cochrane_collaborations_tool_for_assessing.htm. Accessed 03/30, 2016.
- [Background] Henchoz Y, de Goumoens P, Norberg M, Paillex R, So AK. Role of physical exercise in low back pain rehabilitation: a randomized controlled trial of a three-month exercise program in patients who have completed multidisciplinary rehabilitation. Spine (Phila Pa 1976). 2010 May 20;35(12):1192-9. doi: 10.1097/BRS.0b013e3181bf1de9. PMID 20098350
- [Background] Monticone M, Ambrosini E, Rocca B, Magni S, Brivio F, Ferrante S. A multidisciplinary rehabilitation programme improves disability, kinesiophobia and walking ability in subjects with chronic low back pain: results of a randomised controlled pilot study. Eur Spine J. 2014 Oct;23(10):2105-13. doi: 10.1007/s00586-014-3478-5. Epub 2014 Jul 27. PMID 25064093
- [Background] Ostelo RW, Deyo RA, Stratford P, Waddell G, Croft P, Von Korff M, Bouter LM, de Vet HC. Interpreting change scores for pain and functional status in low back pain: towards international consensus regarding minimal important change. Spine (Phila Pa 1976). 2008 Jan 1;33(1):90-4. doi: 10.1097/BRS.0b013e31815e3a10. PMID 18165753
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Hoffmann TC, Glasziou PP, Boutron I, Milne R, Perera R, Moher D, Altman DG, Barbour V, Macdonald H, Johnston M, Lamb SE, Dixon-Woods M, McCulloch P, Wyatt JC, Chan AW, Michie S. Better reporting of interventions: template for intervention description and replication (TIDieR) checklist and guide. BMJ. 2014 Mar 7;348:g1687. doi: 10.1136/bmj.g1687. PMID 24609605
- [Derived] Schmidt AM, Terkildsen Maindal H, Laurberg TB, Schiottz-Christensen B, Ibsen C, Bak Gulstad K, Maribo T. The Sano study: justification and detailed description of a multidisciplinary biopsychosocial rehabilitation programme in patients with chronic low back pain. Clin Rehabil. 2018 Nov;32(11):1431-1439. doi: 10.1177/0269215518780953. Epub 2018 Jun 8. PMID 29879847